CLINICAL TRIAL: NCT01495039
Title: The Role of Oral Nystatin Prophylaxis in ICU Surgical/Trauma Patients
Brief Title: Antifungal Prophylaxis in Intensive Care Unit (ICU) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Filomena Puntillo, Professor, Policlinico Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Nista 1
Record Dates: First submitted 2011-12-12; First posted 2011-12-19 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Fungal Prophylaxis; Candida Infection; Critical Illness; Surgery
MeSH Terms: conditions — Candidiasis; Critical Illness | interventions — Nystatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nystatin (Active Comparator): surgical patients admitted to our ICU older than 18 years of age and expected to require invasive mechanical ventilation for more than 48 h.Patients were allocated to receive systematic nystatin prophylaxis (2 x 106 U per day administered three times daily in the naso-gastric tube)
  Interventions: Drug: Nystatin
- Control (Placebo Comparator): surgical patients admitted to our ICU older than 18 years of age and expected to require invasive mechanical ventilation for more than 48 h.
  Interventions: Drug: Nystatin

INTERVENTIONS:
Drug: Nystatin — Systematic nystatin prophylaxis (2 x 106 U per day administered three times daily in the naso-gastric tube)
  Other Names: Mycostatin

SUMMARY:
Purpose. Oral chemoprophylaxis has been advocated to reduce the incidence of Candida colonization and infection. However, Candida prophylaxis in intensive care unit (ICU) is still a matter of debate.

Methods. Randomized, single-center trial studying single drug (nystatin) versus control in surgical ICU patients. Multiple-site testing for fungi were performed in each patient at ICU admission (T0) and subsequently every 3 days (T3, T6, T9…). The primary evaluation criterion was the time course of colonization index (CI) during ICU stay.

DETAILED DESCRIPTION:
Multiple-site testing for fungi included: tracheal secretions, pharingael swab, stomach contents, rectal swab, groin skin fold swab, urine, and blood. These tests will be performed in each patient at ICU admission (T0) and subsequently every 3 days throughout the ICU stay (T3, T6, T9…), as routine in our ICU.The specimens were placed in a dry medium and taken to the Mycology Laboratory. Group assignment was not indicated on specimens, the mycologists were therefore blinded to treatment allocation.

Each specimen was directly microscopically examined and cultured on Sabouraud media.

ELIGIBILITY:
Inclusion Criteria:

* surgical patients admitted to our ICU older than 18 years of age and expected to require invasive mechanical ventilation for more than 48 h.

Exclusion Criteria:

* pregnancy,
* proven Candida infection,
* prophylactic or curative antifungal treatment within the last 2 months,
* contraindication to oral drug administration,
* known allergy to nystatin or its derivatives, and prior inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
course of the colonization index over time. | AT 15 day from ICU admission
  Fungal colonization will be defined as either the presence of the same yeast on one or more of the six distinct body sites tested (blood sample excepted), or on two consecutive specimens from the same body site. Candida Colonisation index (C.I.)was defined as the ratio of the number of distinct body sites colonised with genotypically identical strains of Candida spp (blood excepted) over the total number of sites tested.

SECONDARY OUTCOMES:
The secondary evaluation criterion will be the occurrence of a fungal infection during the ICU stay | At 15 day from ICU admission
  Fungal infection will be defined as either the presence of a candidemia or the identification of Candida spp. in a normally sterile body site associated with a severe sepsis with negative tests for bacteria or other causes.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bruno, Professor, Study Director — University of Bari; Filomena Puntillo, Professor, Principal Investigator — University of Bari
Locations (1):
- Intensive care Unit, Policlinico Hospital Bari, Bari, Italy, Italy

REFERENCES:
- [Derived] Giglio M, Caggiano G, Dalfino L, Brienza N, Alicino I, Sgobio A, Favale A, Coretti C, Montagna MT, Bruno F, Puntillo F. Oral nystatin prophylaxis in surgical/trauma ICU patients: a randomised clinical trial. Crit Care. 2012 Dec 12;16(2):R57. doi: 10.1186/cc11300. PMID 22490643